CLINICAL TRIAL: NCT04900493
Title: The Rett Syndrome Global Registry
Status: Recruiting | Type: Observational
Sponsor: Rett Syndrome Research Trust (Other)
Collaborators: Baylor College of Medicine (Other); Vanderbilt University Medical Center (Other); Children's Hospital of Philadelphia (Other); Rush University (Other); Boston Children's Hospital (Other); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: Rett-Registry
Record Dates: First submitted 2021-04-26; First posted 2021-05-25 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Rett Syndrome
Keywords: MECP2; Registry; RSRT
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Rett Global Registry is a fully remote, global, caregiver-reported registry to collect information about caring for a loved one with Rett syndrome. In addition, caregivers have the ability to track and graph their loved one's symptoms and care strategies over time, store information for central access, and opt-in to complete medical record consolidation and summary. Qualified researchers and therapeutic developers may request access to de-identified aggregate information to further Rett research, or assist with clinical development planning to facilitate and expedite more effective clinical trials.

DETAILED DESCRIPTION:
The Rett Syndrome Global Registry is a fully remote, global, caregiver-reported registry intended to meet the needs of caregivers, clinicians and researchers, and therapeutic developers with the goal to increase our understanding of this rare disorder, support better outcomes for those with Rett syndrome, and facilitate improved therapeutic development. The Rett Global Registry allows families to provide data about their experience with Rett syndrome to improve their loved one's care while contributing to research. Participants may opt in to track and graph symptoms and care strategies over time to support day-to-day care. Participants may also access aggregate data to see similarities and differences in care strategies and consolidate their personal information in a central location. Participants may opt-in to complete medical record consolidation and summary that is centrally accessible, able to be shared with care providers, and utilized for research.

The registry database is designed and maintained to clinical trial standards and supports research and therapeutic development while meeting or exceeding federal privacy and confidentiality requirements. These datasets including caregiver-reported Rett syndrome progression, quality of life, at home day-to-day data, and consolidated medical records from office visits or hospital stays, provides unique and previously unused sources of information important for improving our understanding of Rett syndrome, allow additional avenues of research, and support therapeutic development. Specifically, the registry is intended to assist with clinical development planning, trial design, trial endpoints, and regulatory filings.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/caregiver must be willing and able to provide written informed consent electronically prior to entering data into the registry.
2. Rett individuals of any age, living or deceased, must have a diagnosis of Rett syndrome and/or have a mutation in MECP2.

Exclusion Criteria:

1. Individuals who have a genetic mutation that is inconsistent with Rett syndrome or who have a different disorder.
2. Individuals with MECP2 Duplication Syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of all ages diagnosed with Rett Syndrome and/or have a mutation in MECP2. MECP2 Duplication syndrome individuals are not included and will be directed to the MECP2 Duplication registries.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of genetic mutation types and clinical diagnoses. | 1 year
  Measured by data obtained from genetic reports and caregiver-reported clinical diagnoses of enrolled patients.
Caregiver report of developmental milestone achievement over time. | 5 years
  Measured by the percent of individuals who have achieved developmental milestones between 1 and 4 times per year.
Caregiver report of symptom burden and development history over time. | 5 years
  Measured by the percent of individuals who report symptoms and their intervention requirements between 1 and 4 times per year.
Caregiver report of composition and frequency of co-morbidities over time. | 5 years
  Measured by the type and number of non-Rett medical conditions between 1 and 4 times per year.
Caregiver report of the composition and frequency of medication and over-the-counter treatments over time. | 5 years
  Measured by the percent of individuals receiving these care strategies by symptom between 1 and 4 times per year.
Caregiver report of the composition and frequency of physician specialty utilization and care received at Rett Clinics over time. | 5 years
  Measured by the type and number of physician specialties used to manage symptoms and the number of individuals who receive care at a Rett clinic between 1 and 2 times per year.
Caregiver report of the composition of the barriers to clinical trial participation over time. | 5 years
  Measured by the type and number of reasons given for individuals not able or willing to participate in clinical trials between 1 and 2 times per year.

SECONDARY OUTCOMES:
Caregiver report of the frequencies of the level of effectiveness for therapies, diets and equipment use over time. | 5 years
  Measured by percent of patients perceiving these care strategies as successful between 1 and 2 times per year.
Caregiver report of the frequencies of the level of effectiveness, degree of side effect severity, and other symptom impacts of medications and over-the-counter treatments over time. | 5 years
  Measured by percent of patients receiving medications or over-the-counter treatments and the percent perceiving these care strategies as successful, with side effects, and impact on other symptoms between 1 and 4 times per year.
Caregiver report of the percent of individuals requiring emergency care and unplanned hospital admissions over time. | 5 years
  Measured by the number of patients requiring emergency care and hospital admissions at least 1 time per year.
Percent of individuals using registry features, including tracking, medical record consolidation, central storage, and family connections over time. | 5 years
  Measured by the number of individuals using these features between 1 and 4 times per year.

OTHER OUTCOMES:
Number of research studies conducted through the registry for the purpose of collecting new data over time. | 5 years
  Measured by the number of studies initiated at least 1 time per year.
Number of research studies conducted with existing datasets for the purpose of mining registry data over time. | 5 years
  Measured by the number of studies initiated at least 1 time per year.

CONTACTS AND LOCATIONS:
Overall Officials: Jana von Hehn, PhD, Principal Investigator — Rett Syndrome Research Trust
Locations (1):
- Rett Syndrome Research Trust, Trumbull, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified Investigators may make data requests to the Rett Syndrome Global Registry Oversight Committee
Supporting Information: ICF
Time Frame: Data will be available upon achieving a threshold enrollment of 500 participants.
Access Criteria: Qualified Investigators interested in advancing Rett Syndrome research or therapeutic development.